CLINICAL TRIAL: NCT04366102
Title: Multisensory Stimulation and Soft Tissue Therapy on Procedural Pain and Neurodevelopment Among Preterm Neonates (MUST-P3) Randomized Controlled Trial
Brief Title: Reducing Pain and Promoting Neurodevelopment Among Preterm Neonates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asir John Samuel (Other)
Collaborators: Department of Science and Technology, Government of India (Unknown); Maharishi Markendeswar University (Deemed to be University) (Other)
Responsible Party: Sponsor-Investigator, Asir John Samuel, Associate professor, Maharishi Markendeswar University (Deemed to be University)
Organization: Maharishi Markendeswar University (Deemed to be University) (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MMDU/IEC/2152; U1111-1242-9663 (Other: Universal Trial Number (UTN)-WHO)
Record Dates: First submitted 2020-04-25; First posted 2020-04-28 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Neonatal Disease; Neonatal Disorder
Keywords: Neonates; Pain
MeSH Terms: conditions — Infant, Newborn, Diseases; Pain | interventions — Therapy, Soft Tissue

STUDY DESIGN:
Intervention Model Description: Neonates admitted in the Neonatal intensive care unit will be divided randomly into 2 groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Multisensory stimulation and soft tissue therapy
  Interventions: Other: Multisensory stimulation with soft tissue therapy
- Group B (Experimental): Routine Hospital care
  Interventions: Other: Routine hospital care

INTERVENTIONS:
Other: Multisensory stimulation with soft tissue therapy — Multisensory stimulation with soft tissue therapy will be given. Multisensory stimulation consists of Auditory, vestibular, tactile, olfactive, oromotor, Visual, and Kinesthetic stimulation. Soft tissue therapy consists of stroking, effleurage, fingertip kneading, tapping, and skin rolling will be given. Total intervention will be given for 30 min. 5 times per week
  Arms: Group A
Other: Routine hospital care — Routine hospital care will be given to the preterm neonates
  Arms: Group B

SUMMARY:
To determine the effects of multisensory stimulation and soft tissue therapy on procedural pain and neurodevelopment among neonates admitted to the NICU is the aim of the study. The study will be two groups randomized clinical trial of five days intervention program. The intervention will be given among two groups. Group A will receive both multisensory stimulation and soft tissue therapy, Group B will receive only regular hospital care. The PIPP and N-PASS will be used for assessing pain. The INFANIB and Premie-Neuro will be used for assessing neuromotor development among neonates. The outcomes will be taken before and after the fifth day of the intervention. Multisensory stimulation and soft tissue therapy might help in reducing pain and promoting neurodevelopment.

DETAILED DESCRIPTION:
This study will utilize two parallel groups, randomised design to analyze the effects of soft tissue therapy and multisensory stimulation on pain and neurodevelopment. 104 neonates admitted in NICU will be recruited through purposive sampling for the trial. Procedural pain will be assessed with PIPP and N-PASS through recorded video. Neurodevelopmental outcomes will be assessed with INFANIB Scale and Premie-Neuro. The measurements will be taken after 24 hours of birth at the baseline and after the fifth day of the intervention. The treatment will be given into two groups i.e. Group A (Multisensory stimulation and soft tissue therapy group), Group B (routine hospital care). MSS will consist of Auditory Stimulation, Tacto-Kinesthetic stimulation, Vestibular stimulation, Visual stimulation, Oral-stimulation, and Olfactive stimulation. Soft tissue therapy consisted of stroking, effleurage, skin rolling, and kneading techniques, Will be given in 5 Phases-Forehead and face, Back and Neck, Chest and abdomen, upper-lower limbs. Total 30 min. of the treatment plan, per day, will be given to the neonates, after 30 min. of feed, for up to 5 days of NICU stay.

ELIGIBILITY:
Inclusion Criteria

* Preterm between 30- 36 weeks of gestation
* Birth weight >1000 g
* Not receiving analgesics/sedatives
* APGAR score ranged between 4-6 in 1 min. & 7 to 9 in 5 min.
* Undergoing routine healthcare procedures in NICU

Exclusion Criteria

* Preterm with surgery
* Preterm having unstable vitals
* Preterm with congenital malformations
* Preterm who require mechanical ventilation
* Having inborn errors of metabolism and also with seizures disorders,

Ages: 24 Hours to 5 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 68 (Actual)
Dates: Start 2020-10-22 (Actual); Primary Completion 2023-09-16 (Actual); Study Completion 2023-10-20 (Actual)

PRIMARY OUTCOMES:
The Premature infant pain profile-Revised (PIPP-R) | Change score of PIPP at the baseline(immediately after painful procedure, at 30s, 60s, 90s, and 120s) and after five days of intervention
  Measuring procedural pain among neonates, having 1 to 3 scoring. 0 describe normal and 3 describes low score
Neonatal pain agitation sedation scale (N-PASS) | Change score of N-PASS at the baseline(immediately after painful procedure, at 30s, 60s, 90s, and 120s) and after five days of intervention
  Measuring procedural pain along with sedation, having score ranged from 0 to 2, 0 describes normal and 2 describes low score

SECONDARY OUTCOMES:
Infant neurological international battery (INFANIB) | Change score of INFANIB at the baseline and after five days of intervention
  Measuring neurodevelopmental outcomes among preterm neonates. Scoring is from 5, 3, and 1. Score 5 means Normal, score 3 means mildly abnormal, score 1 means markedly abnormal. Total score for preterm neonate is 70.
Premie-Neuro | Change score of Premie-Neuro at the baseline and after five days of intervention
  Premie-neuro used for measuring neurodevelopmental outcome in preterm neonates between 23 and 37 weeks of gestation. It has total 24 items. Each item has a score of 1,3, and 5. Total score is 120. Score less than 70 is considered as abnormal, score between 70-99 is questionable, and score above 100 is normal.

CONTACTS AND LOCATIONS:
Overall Officials: Neha Sharma, MPT, Principal Investigator — Maharishi Markandeshwar institute of Physiotherapy and Rehabilitation; Asir J Samuel, MPT, PhD, Study Chair — Maharishi Markandeshwar Institute of physiotherapy and Rehabilitation; Kusum Mahajan, MD, Study Chair — Maharishi Markandeshwar Institute of Medical Sciences & Research
Locations (1):
- Neonatal Intensive Care Unit, Maharishi Markandeshwar Hospital, Ambāla, Haryana, India

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) will be shared via Mendeley Dataset
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Study Protocol - December, 2020 Statistical Analysis Plan (SAP) - December, 2020 Informed Consent Form (ICF) - December, 2020
Access Criteria: By publishing study protocol with detailed statistical Analysis Plan in SCOPUS and PubMed indexed journals

REFERENCES:
- [Background] Zeraati H, Nasimi F, Rezaeian A, Shahinfar J, Ghorban Zade M. Effect of Multi-sensory Stimulation on Neuromuscular Development of Premature Infants: A Randomized Clinical Trial. Iran J Child Neurol. 2018 Summer;12(3):32-39. PMID 30026767
- [Background] de Melo GM, Lelis AL, de Moura AF, Cardoso MV, da Silva VM. [Pain assessment scales in newborns: integrative review]. Rev Paul Pediatr. 2014 Dec;32(4):395-402. doi: 10.1016/j.rpped.2014.04.007. PMID 25511005
- [Derived] Sharma N, Samuel AJ. Multisensory Stimulation and Soft Tissue Therapy on Pain and Neurodevelopment Among Preterm Neonates. Pediatr Phys Ther. 2022 Apr 1;34(2):277-282. doi: 10.1097/PEP.0000000000000887. PMID 35385466
- See also: Effect of Multi-sensory Stimulation on Neuromuscular Development of Premature Infants: A Randomized Clinical Trial — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC6045934/
- See also: Pain assessment scales in newborns: integrative review — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4311795/